CLINICAL TRIAL: NCT03420040
Title: A Comparative Study of the Effects of QS-M Needle Free Injector and Glargine Pen Subcutaneous Injection of Insulin Glargine on Insulin Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: KY20172077-1
Record Dates: First submitted 2018-01-09; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glargine Insulin; QS-M Needle Free Injector
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QS-M Needle Free Injector group (Experimental): To observe the use of insulin in glycemia under good blood glucose control in the QS-M Needle Free Injector group.
  Interventions: Device: QS-M Needle Free Injector
- Glargine pen group (Active Comparator): To observe the amount of insulin used by the Glargine pen group under good blood glucose control.
  Interventions: Device: Glargine pen

INTERVENTIONS:
Device: QS-M Needle Free Injector — The subjects were proficient in the two injection methods of injection of QS-M needle free syringe and Glargine pen injection
  Arms: QS-M Needle Free Injector group
Device: Glargine pen — The subjects were proficient in the two injection methods of injection of QS-M needle free syringe and Glargine pen injection
  Arms: Glargine pen group

SUMMARY:
A clinical study of the use of glargine insulin in 2 subjects with type two diabetes in China was carried out. The two kinds of injection methods were evaluated as subcutaneous injection of insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

1. male or female aged 18-70 years of age, women of childbearing age need to take adequate contraceptive measures to minimize the risk of pregnancy;
2. the standard of diagnosis of type 2 diabetes and the course of the disease is more than half a year;
3. 18 Kg/m2 = BMI = 30Kg/m2;
4. received daily injections of insulin glargine and also take one to three kinds of oral medicine (not including secretagogues) patients, daily insulin glargine total dose more than 12IU but <50IU, the use of insulin glargine than in January;
5. the blood glucose in the fasting vein was in 5.0-9.0mmol/L;
6. the letter of informed consent has been read and signed.

Exclusion Criteria:

1. there is conflict of interest with this research.
2. blood glucose control is not good enough to participate in this study, such as repeated hypoglycemia, diabetic ketoacidosis or hyperosmolar coma.
3. serious diabetic complications such as diabetic foot, diabetic nephropathy and so on;
4. severe cardiovascular events occurred in the last 6 months.
5. the application of hormone or immunosuppressant, or low immunity defect;
6. the use of non steroidal anti-inflammatory drugs;
7. the use of sulfonylureas and insulin secreting agents;
8. a person with a history of cancer;
9. a history of unstable or rapid progressive renal disease;
10. an unstable history of major mental illness;
11. the history of hemoglobin (such as sickle red cell anemia, thalassemia, iron granulocytic anemia);
12. women who are pregnant or are breastfeeding;
13. in the near future there is a clear infection, such as urinary tract infection and pneumonia;
14. recent important visceral hemorrhage, such as gastric hemorrhage and cerebral hemorrhage, etc.
15. skin diseases such as exfoliative dermatitis, pustular sore and infection of pyogenic bacteria;
16. the history of acute pancreatitis or pancreatectomy;
17. the researchers believe that it may lead to any situation in which the subject is unable to complete the study or may cause significant risk to the subject.
18. the results of the laboratory examination are as follows: A. obvious abnormal liver function or in the active phase of the disease (AST> 3 times the upper limit of normal ALT> or 3 times the upper limit of normal); The creatinine clearance rate of B. was <60ml/min; C. anaemia caused by any cause of the disease; The results of pregnancy test in women of childbearing age of D. were positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-02-20 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in fasting blood glucose between baseline to week 4 | baseline and week 4
  fasting blood glucose are measured at baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Qiuhe Ph.D Ji, M.D., Principal Investigator — Department of Endocrinology, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Xijing Hospital, Fourth Military Medical university, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Xing Y, Xie X, Xu J, Liu J, He Q, Yang W, Zhang N, Li X, Wang L, Fu J, Zhou J, Gao B, Ming J, Liu X, Lai J, Liu T, Shi M, Ji Q. Efficacy and safety of a needle-free injector in Chinese patients with type 2 diabetes mellitus treated with basal insulin: a multicentre, prospective, randomised, crossover study. Expert Opin Drug Deliv. 2019 Sep;16(9):995-1002. doi: 10.1080/17425247.2019.1649251. Epub 2019 Aug 5. PMID 31359813